CLINICAL TRIAL: NCT05924399
Title: Affect Labeling: A Promising New Approach for Mitigating PTSD
Brief Title: PTSD Affect Labeling Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Defense Group, Inc. (Unknown); Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Craske, Co-Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: W911NF-14-C-0056
Record Dates: First submitted 2023-06-06; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Post-traumatic Stress Disorder; Post-Traumatic Stress Disorder, Chronic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Affect Labeling Training (Experimental): Participants complete a total of six training sessions, twice a week for three consecutive weeks. In each session, they spend 40 minutes completing computer-based inhibitory regulation training utilizing four strategies.
  Interventions: Behavioral: Affect Labeling Training

INTERVENTIONS:
Behavioral: Affect Labeling Training — (1) Participants will view combat-relevant images and then label the image or how they feel while viewing the image. (2) Participants will view facial expressions and then label the image. (3) Participants will view negative combat- irrelevant images (such as snakes or spiders) and then label the image or how they feel while viewing the image. (4) Participants will complete Go-NoGo trials similar to the fMRI Go-NoGo task described above. Participants will receive all four types of inhibitory training.

SUMMARY:
The overall goal of this study is to use fMRI and psychophysiological measures to investigate a novel strategy involving "Affect Labeling" for improving emotion regulation in PTSD that could lead to a new treatment regimen for PTSD.

Our project has two specific aims. First, the investigators aim to identify a novel neural target for possible PTSD intervention by verifying that RVLPFC-based inhibitory processing is impaired in PTSD. Second, the investigators will examine whether repeated practice with a simple cognitive-emotional task that requires inhibitory processing, namely, affect labeling, can strengthen the RVLPFC's ability to down-regulate emotional responses and physiological reactivity in PTSD and thereby form the basis of a novel treatment strategy to be developed in future studies. Secondary objectives are to examine the extent to which RVLPFC-based inhibitory impairments in PTSD are specific to trauma-relevant emotional processing (i.e., trauma-related distress) or extend to other types of inhibitory regulation in general, which would have implications for the future study of inhibitory-enhancement-based interventions for PTSD.

DETAILED DESCRIPTION:
Previous research suggests that individuals with PTSD have impaired RVLPFC- based inhibitory regulation. Such deficits would appear to contribute to poor inhibitory regulation of emotional responses when faced with trauma-reminders, which represents a core pathological mechanism of PTSD.

However, no previous studies have directly examined RVLPFC-based inhibitory deficits of emotional responses in PTSD. Affect labeling is a simple process that involves linguistic processing of emotional responses, for example, verbally labeling current feelings as "anxious" or "angry", and is an established form of affective inhibitory regulation involving RVLPFC down-regulation of amygdala-based affective responses. Therefore, the investigators will test whether PTSD is associated with impaired RVLPFC-based emotional inhibitory processing compared to healthy control participants by performing fMRI scan while they use affect labeling to label their own emotional responses to emotionally-evocative images relevant to their trauma. The investigators will then test whether repeated practice with affect labeling will "repair" the impaired RVLPFC inhibitory control in PTSD, by strengthening the capacity of the RVLPFC to down-regulate amygdala responses. In support of this idea, the investigators have previously demonstrated that exposure therapy augmented with affect labeling was more effective in reducing fear responses than exposure alone in specific phobia (Kircanski et al., 2013). In the present study, following the initial baseline fMRI scan mentioned above, participants with PTSD will complete three weeks of affect labeling training and then undergo a second fMRI scan to again assess inhibitory regulation capacity.

The investigators hypothesize that, compared to healthy (without PTSD) subjects, participants with PTSD will exhibit less RVLPFC activity, more amygdala activity (i.e., less amygdala deactivation), as well as less inverse correlation between the RVLPFC and the amygdala at baseline, reflecting impaired inhibitory regulation. In addition, the investigators hypothesize that participants will exhibit increased physiological reactivity compared to healthy control subjects.

The investigators also hypothesize that affect labeling training will lead to increased inhibitory regulation success, which will be reflected by increased RVLPFC activity, decreased amygdala activity, increased inverse connectivity between RVLPFC and amygdala from pre to post training. The results from this initial effort will form the foundation for future studies examining affect labeling training as a bona fide treatment strategy for PTSD.

ELIGIBILITY:
INCLUSION CRITERIA

Inclusion Criteria for All Veteran Participants (Ps):

1. All Ps must be veterans with deployment experience.
2. Ps must meet DSM-IV criterion "A" for PTSD, which requires exposure to a traumatic event involving actual or threatened physical injury or death. This trauma must have occurred during military service, but may take a variety of forms (e.g., injury to self, witnessing death of another, etc.).
3. Ps must be 18-45 years old (18-60 for non-fMRI Ps) since normal age-related structural and functional variations in participants above and below this age range could prevent accurate comparison of neural activity across participants.
4. Ps must be English-speaking as translation of all study materials into other languages would be cost-prohibitive.
5. Both male and female participants are allowed.
6. Ps who will complete the fMRI must be right-handed in order to allow comparison of neural activity across participants.

Additional Inclusion Criterion for PTSD Participants (PTSDs): PTSDs must meet full DSM- IV criteria for PTSD with a trauma related to their military service, as assessed by the CAPS.

Additional Inclusion Criterion for Healthy Control Participants (HCs): HCs must not meet DSM-IV criteria for current/lifetime PTSD or any other current Axis I disorders.

Inclusion Criteria for Non-Veteran Healthy Controls:

1. Must be 18-45 years old
2. Must be English-speaking
3. Male or female participants are allowed

EXCLUSION CRITERIA

Exclusion Criteria for All fMRI Participants:

1. Ps must not have any metallic implants or other non-removable metal in the body (e.g., shrapnel, surgical staples or screws, etc.) as this would preclude them from undergoing any MRI scanning.
2. Ps must not be claustrophobic in order to be able to complete all fMRI procedures.
3. Ps must not be pregnant (as assessed by verbal report) as the research question is not pregnancy-related.
4. Ps must not have any serious unstable medical illnesses.
5. Ps must not have intellectual impairment, bipolar disorder, psychosis, delusional disorder, or suicidality.
6. Ps must not have any organic brain damage, including a history of moderate to severe traumatic brain injury (TBI), as this would confound analyses comparing activations across subjects. A history of mild TBI is allowed.
7. Ps must not meet DSM-IV criteria for Substance Dependence within the last six months due to both the possibility of neural changes associated with the substance use, and issues of participant safety.
8. Ps must not have made any recent modifications to psychotropic medication status (i.e., within the last 1 month for benzodiazepines and within the last 3 months for SSRI and SSNIs).
9. Ps must not have recently initiated or made changes to any psychotherapy (within the last 3 months).
10. Ps must not have had any chronic or repeated neglect/maltreatment, sexual abuse, physical abuse, emotional abuse, or domestic violence prior to the age of 7 (as assessed with the Early Trauma Inventory and CAPS), given evidence for adverse brain development and structural abnormalities in this subgroup of individuals.

Exclusion Criteria for All Non-fMRI Participants:

1. Ps must not be pregnant (as assessed by verbal report) as the research question is not pregnancy-related.
2. Ps must not have any serious unstable medical illnesses.
3. Ps must not have intellectual impairment, bipolar disorder, psychosis, delusional disorder, or suicidality.
4. Ps must not meet DSM-IV criteria for Substance Dependence within the last six months due to issues of participant safety.
5. Ps must not have made any recent modifications to psychotropic medication status (i.e., within the last 1 month for benzodiazepines and within the last 3 months for SSRI and SSNIs).
6. Ps must not have recently initiated or made changes to any psychotherapy (within the last 3 months).

Additional Exclusion Criterion for PTSD Participants (PTSDs):

The investigators will exclude highly-dissociative individuals, defined as those who score 15 or higher on the Clinician Administered Dissociative States Scale (Bremner et al., 1998). While the majority (i.e., 70%) of individuals with PTSD are characterized by prefrontal under-regulation and limbic over-responding to trauma cues, research has also identified a subgroup of PTSD individuals, up to 30%, who are characterized as highly 'dissociative' and exhibit the opposite neural pattern to trauma cues, i.e., abnormally low and over-regulated amygdala responses (Lanius et al., 2010). The current proposal focuses on the former, larger group of less-dissociation-prone PTSD individuals with inhibitory deficits, as this appears to be the group for whom inhibitory enhancement may be particularly helpful. Accordingly, the investigators will exclude those with high levels of baseline dissociative symptomology in this first proof-of-concept study.

Exclusion Criteria for Non-Veteran Healthy Controls:

1. Ps must not have been exposed to a DSM-IV defined traumatic event.
2. Ps must not meet criteria for any current DSM-IV Axis I disorder and must not have intellectual impairment or current suicidality.
3. Ps must not be pregnant (as assessed by verbal report) as the research question is not pregnancy-related.
4. Ps must not have any serious unstable medical illnesses.
5. Ps must not be currently receiving treatment for a psychiatric problem (including psychotherapy and psychotropic medication).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2015-10-09 (Actual); Study Completion 2015-10-09 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affective Schedules - State & Trait Versions (PANAS) | Change from baseline to Post-AL Training (3 weeks from baseline)
  The PANAS is a widely used measure comprising 20-items assessing activated forms of Positive Affect and Negative Affect using 5-point scales (1 = very slightly/not at all, 5 = extremely). Higher scores on each subscale (positive affect and negative affect) reflect higher levels of positive and negative affect, respectively.
Mood and Anxiety Symptom Questionnaire - Mini Version | Change from baseline to Post-AL Training (3 weeks from baseline)
  The Mini-MASQ is a 26-item measure of mood and anxiety symptoms developed to evaluate predictions of the tripartite model of anxiety and depression. The MASQ has three subscales: (1) General Distress (GD: 8 items), (2) Anxious Arousal (AA: 10 items), and (3) Anhedonic Depression (AD: 8 items). Respondents indicate the extent to which they experienced each symptom during the past week from 1=not at all to 5=extremely.
Emotion Regulation Questionnaires (ERQ) | Change from baseline to Post-AL Training (3 weeks from baseline)
  The ERQ is a 10-item measure designed to assess individual differences in the habitual use of two emotion regulation strategies: cognitive reappraisal and expressive suppression.
fMRI Inhibitory regulation of trauma-relevant emotion | Change from baseline to Post-AL Training (3 weeks from baseline)
  The primary outcome variables for our key objectives will be neural activity obtained during the baseline fMRI scans for participants with PTSD (PTSDs) vs. healthy controls (HCs) as well as changes in neural activity from pre to post training for PTSDs.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Change from baseline to Post-AL Training (3 weeks from baseline)
  Clinician-reported PTSD symptom severity
Mindful Attention Awareness Scale (MAAS) | Change from baseline to Post-AL Training (3 weeks from baseline)
  The trait MAAS is a 15-item scale designed to assess a core characteristic of mindfulness, namely, a receptive state of mind in which attention, informed by a sensitive awareness of what is occurring in the present, simply observes what is taking place.
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to Post-AL Training (3 weeks from baseline)
  Self-reported PTSD symptom severity. The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD using a 5-point Likert scale of how much they were bothered by each symptom (0 = "not at all" to 4 = "extremely"). Scores are summed and higher scores represent greater self-reported PTSD symptoms. Scores range from 0-80.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Burklund, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Burklund LJ, Davies CD, Niles A, Torre JB, Brown L, Vinograd M, Lieberman MD, Craske MG. Affect labeling: a promising new neuroscience-based approach to treating combat-related PTSD in veterans. Front Psychol. 2024 Jun 7;15:1270424. doi: 10.3389/fpsyg.2024.1270424. eCollection 2024. PMID 38911954